CLINICAL TRIAL: NCT00588198
Title: Study of Peripheral Blood and/or Bone Marrow, Including Detection of Occult Metastases, in Patients With Melanoma
Brief Title: Peripheral Blood and/or Bone Marrow, Including Detection of Occult Metastases, in Patients With Melanoma
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 91-125
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Melanoma
Keywords: histologically confirmed melanoma of any site
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Melanoma patients

SUMMARY:
The purpose of this study is to determine if tumor cells can be detected in the peripheral blood and/or bone marrow of patients with melanoma.

DETAILED DESCRIPTION:
Patients with melanoma can succumb to subclinical metastatic disease, not detectable at presentation by conventional physical examination, hematologic and biochemical screening, or radiologic evaluation. More intensive radiologic evaluation with CT or radioisotope scanning has not proven to be useful. What may be useful is a more sensitive method of staging melanoma patients at presentation, specifically evaluating them for subclinical systemic disease.

ELIGIBILITY:
Inclusion Criteria:

MSK Patients with histologically confirmed melanoma of any site and at least one of the following:

* Primary tumor > 4.0 mm thick (AJCC Stage IIB)
* Clinically or histologically positive regional nodes (AJCC Stage III)
* Any in transit disease (AJCC Stage III)
* Any systemic metastases (AJCC Stage IV)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Melanoma Patients seen at Memorial Sloan-Kettering Cancer Center (MSK)
Sampling Method: Non-Probability Sample
Enrollment: 754 (Actual)
Dates: Start 1991-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Assess the sensitivity of RT-PCR to detect evidence of melanoma cells in bone marrow and/or peripheral blood and estimate sensitivity separately for each of the different stage groupings for melanoma | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Danile Coit, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org